CLINICAL TRIAL: NCT01198691
Title: Closure of Pfannenstiel Skin Incisions After Cesarean Delivery: A Comparison of Metallic Staples Versus Absorbable Staples
Brief Title: A Comparison of Metallic Staples Versus Absorbable Staples After a Cesarean Section (C-Section)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10018-10-016
Record Dates: First submitted 2010-09-02; First posted 2010-09-10 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2014-05

CONDITIONS: Cesarean Section
Keywords: metallic staples; absorbable staples; Cesarean Delivery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): This group will receive the standard metallic staples to close their incision.
  Interventions: Device: Insorb absorbable staples
- Case Group (Experimental): This group will receive the Insorb absorbable staples to close their incision.
  Interventions: Device: Insorb

INTERVENTIONS:
Device: Insorb absorbable staples — Patients will be randomized to receive either the standard metallic staples or the Insorb absorbable staples
  Arms: Control Group
Device: Insorb — Patients will be randomized to receive either standard metallic staples or Insorb absorbable staples
  Arms: Case Group

SUMMARY:
The purpose of the study is to compare post operative pain, cost effectiveness, speed of closure and patient satisfaction of Pfannenstiel incisions closed with metallic staples versus absorbable staples (Insorb) after Cesarean Delivery.

DETAILED DESCRIPTION:
The ideal method of closing the skin following a Pfannenstiel incision has not yet been established. Presently, the method of skin closure is a matter of the surgeon's personal preference. Currently, there is limited evidence regarding which method is considered "superior" in terms of post operative pain, patient satisfaction, and cost effectiveness. This information would be incredibly valuable in helping guide surgeons in their choice of skin closure technique; and with the rates of Cesarean deliveries rapidly rising, it is important to determine the best method of skin closure in order to optimize patient care.

After a patient is consented she will be randomized into either the control group and receive the standard metallic staples or the experimental group and receive the absorbable staples for her skin closure procedure. One day after her procedure the RN will ask the patient to rate her pain using a 10cm VAS pain scale. Two or three days after the skin closure and before the patient is discharged a short survey about the patient's satisfaction of her scar appearance will be administered. The PI will go back and review the patient's chart to determine the amount of narcotics administered.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric service patients (receiving prenatal care from the Faculty Medical Center)
* Women greater than 18 years old
* Singleton gestation
* Cesarean Section performed by Pfannenstiel skin incision

Exclusion Criteria:

* History of drug or alcohol abuse
* Contraindication to post operative NSAID's or Narcotics
* Emergent Cesarean Deliveries
* Less then 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Feese CA, Johnson S, Jones E, Lambers DS. A randomized trial comparing metallic and absorbable staples for closure of a Pfannenstiel incision for cesarean delivery. Am J Obstet Gynecol. 2013 Dec;209(6):556.e1-5. doi: 10.1016/j.ajog.2013.08.001. Epub 2013 Aug 3. PMID 23921089

RESULTS

PARTICIPANT FLOW:
Period: Completed Surgery -Received Intervention
Arm/Group | Control Group | Case Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Completed VAS Score Postop Day 1
Arm/Group | Control Group | Case Group
Started | 50 | 50
Completed | 47 | 46
Not Completed | 3 | 4
Period: Completed VAS Score at Discharge
Arm/Group | Control Group | Case Group
Started | 50 (Missing a VAS score on postop day one did not exclude participants from having a score at discharge.) | 50 (Missing a VAS score on postop day one did not exclude participants from having a score at discharge.)
Completed | 45 | 44
Not Completed | 5 | 6
Period: Survey Prior to Discharge
Arm/Group | Control Group | Case Group
Started | 50 (Survey was given to all participants even if they were missing data from previous periods.) | 50 (Survey was given to all participants even if they were missing data from previous periods.)
Completed | 18 | 17
Not Completed | 32 | 33
Period: 6 Week Post-partum Survey
Arm/Group | Control Group | Case Group
Started | 50 (Survey was sent to all participants even if they were missing data from the previous two periods.) | 50 (Survey was sent to all participants even if they were missing data from the previous two periods.)
Completed | 21 | 26
Not Completed | 29 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Case Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.32 (5.63) | 27.38 (6.15) | 27.85 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | 22 | 23 | 45
  White/Caucasian | 24 | 26 | 50
  Asian | 2 | 0 | 2
  Pacific Islander | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain
Description: Post operative pain at post operative day #1 will be measured using the Visual Analogue Scale (VAS). The scale has a minimum score of 0 representing no pain and a maximum score of 10 representing the worst possible pain.
Time Frame: 1 Year
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 47 | 46
units on a scale | 2.56 (1.47) | 2.90 (1.54)

2. Primary Outcome: Post Operative Pain (3 Days Post-op)
Description: Post operative pain at the time of discharge will be measured using the Visual Analogue Scale (VAS). The scale has a minimum score of 0 representing no pain and a maximum score of 10 representing the worst possible pain.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 45 | 44
units on a scale | 2.66 (1.47) | 3.52 (5.80)

3. Secondary Outcome: Patient Satisfaction
Description: Patients will be given a survey prior to being discharged to assess their satisfaction with the appearance of their scar. The survey asked whether patients "strongly agree," "agree," "disagree," or "strongly disagree" with the statement, "I am satisfied with the overall appearance of my incision." Those who responsed "agree" or "strongly agree" were said to be satisfied with the appearance and the outcome is reported as number of participants who were satisfied.
Time Frame: This will be assessed 3 day after the patient's C-section before they are discharged from the hospital
Measure: Number; unit: participants
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 18 | 17
participants | 16 | 14

4. Secondary Outcome: Patient Satisfaction
Description: Patients will be given a survey at their 6 week post-op visit to assess their satisfaction with the appearance of their scar. The survey asked whether patients "strongly agree," "agree," "disagree," or "strongly disagree" with the statement, "I am satisfied with the overall appearance of my incision." Those who responsed "agree" or "strongly agree" were said to be satisfied with the appearance and the outcome is reported as number of participants who were satisfied.
Time Frame: Patient satisfaction will be assessed 6 weeks later at their post-op visit
Measure: Number; unit: participants
Arm/Group | Control Group | Case Group
Number analyzed (Participants) | 21 | 26
participants | 20 | 21

ADVERSE EVENTS:
Time Frame: Duration of study: July 2010 - May 2011 (10 months).
Arm/Group | Control Group | Case Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Low response rate to patient surveys at discharge and at 6 weeks postpartum.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes